CLINICAL TRIAL: NCT02458677
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study of PRX003 Administered by Intravenous Infusion in Healthy Subjects
Brief Title: Single Ascending Dose Study of PRX003 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prothena Biosciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRX003-CL001
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRX003 (Experimental)
  Interventions: Drug: PRX003
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PRX003
  Arms: PRX003
Other: Placebo
  Arms: Placebo

SUMMARY:
This single ascending dose study is to determine safety, tolerability, pharmacokinetics and immunogenicity of PRX003 in approximately 40 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Body mass index (BMI) between 18-32 kg/m2 with a minimum weight of 45 kg
* Female subjects must be surgically sterile or post-menopausal or if of child-bearing potential must use contraception
* Male subjects and their partners of childbearing potential must use contraception

Exclusion Criteria:

* Positive test for drug of abuse
* Past or current history of alcohol abuse
* Positive for TB, hepatitis B, hepatitis C or HIV infection

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as determined by number of subjects with adverse events | Up to 3 months
Determination of pharmacokinetics parameters-(Cmax) | Up to 3 months
  maximum concentration (Cmax)
Determination of pharmacokinetics parameters-(AUClast) | Up to 3 months
  area under the concentration-time curve from time zero to the last quantifiable concentration time-point (AUClast)
Determination of pharmacokinetics parameters-(AUCinf) | Up to 3 months
  area under the concentration-time curve from time zero extrapolated to infinity (AUCinf)
Determination of pharmacokinetics parameters-elimination rate constant | Up to 3 months
  elimination rate constant
Determination of pharmacokinetics parameters-(t½) | Up to 3 months
  terminal elimination half life (t½)
Determination of pharmacokinetics parameters-(CL) | Up to 3 months
  clearance (CL)
Determination of pharmacokinetics parameters-(Vd) | Up to 3 months
  apparent volume of distribution (Vd)

SECONDARY OUTCOMES:
Immunogenicity as determined by measurement of anti-PRX003 antibodies | Up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials Early Phase Services, San Antonio, Texas, United States